CLINICAL TRIAL: NCT03590535
Title: Fifth Generation Cardiac Troponin-T (cTnT) Assays in Emergency Department (ED) Evaluation of Possible Acute Coronary Syndromes (ACS)
Brief Title: 5th Generation cTnT in ED ACS
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAAR7939
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Emergency Department (ED)
MeSH Terms: conditions — Acute Coronary Syndrome; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Possible ACS: Adult patients presenting to the Emergency Department with symptoms that maybe be caused by acute coronary syndrome, who are clinically considered to be at enough risk for ACS to send a cardiac enzyme as part of the diagnostic evaluation.
  Interventions: Diagnostic Test: 4th Gen cTnT; Diagnostic Test: 5th Gen cTnT

INTERVENTIONS:
Diagnostic Test: 4th Gen cTnT — Current "Fourth" Generation Cardiac Troponin T Enzyme Assay
  Other Names: cTnT; cardiac troponin-T
Diagnostic Test: 5th Gen cTnT — New "Fifth" Generation ("High-sensitivity") Troponin T Enzyme Assay
  Other Names: hs-cTnT; high-sensitivity cardiac troponin-T

SUMMARY:
This study intends to investigate the usefulness of the new "5th generation" cardiac troponin enzyme in determining which patients presenting with possible acute coronary syndrome can be quickly and safely discharged or admitted from the Emergency Department. The investigators hypothesize that introducing this enzyme into practice will reduce the time it takes to make decisions about admitting or discharging these patients with no increase in adverse events in the discharged patients.

DETAILED DESCRIPTION:
The workup of patients for acute coronary syndrome (ACS) is one of the most common diagnostic considerations in medicine today. Chest pain is the cause of over 7 million annual emergency visits in the United States alone, representing over $10 billion in annual healthcare costs. Because of the significant morbidity and mortality associated with ACS, as well as the perception that there is a greater degree of professional liability associated with its misdiagnosis, a disproportionate amount of clinical energy and resources are currently employed to either make ("rule-in") or exclude ("rule-out") the diagnoses. Yet only a small fraction of these patients are eventually diagnosed with ACS. The combination of high importance paired with significant clinical heterogeneity makes it a diagnosis that is made with great difficulty and at great expense.

For the past several decades serial measurements of cardiac biomarkers over a period of several hours have been the mainstay of ACS evaluation. More recently, "high sensitivity" assays for the troponin enzyme, the most widely followed marker of cardiac injury, have been introduced for clinical use outside of the United States.

These high-sensitivity cardiac troponin (hs-cTn) assays have been shown to be more sensitive for detecting injury to cardiac myocytes and have been employed in protocols that allow for a more rapid rule-in and rule-out of ACS in European, Canadian, and Australasian settings. In 2017, the FDA approved the Roche Elecsys Troponin T Gen 5 Stat (5th Gen Tn) assay for clinical use in the United States.

The American medical community has responded to this with both eagerness and trepidation. Despite large clinical trials demonstrating the utility of these new assays in study populations, it is unclear what the impact will be on clinical practice. There is an understandable concern among providers that this highly sensitive assay will identify many patients with elevated levels of troponin from non-ACS causes and with uncertain clinical significance. There is also uncertainty because studies performed in European populations may not be applicable to the multi-ethnic populations that present to US emergency departments.

While there is much literature that attests to the performance of the test in study settings, there is less understanding of the impact of this assay on real-world practice settings. Therefore, it is critically important that we track and study how the new assay affects provider practice and clinical outcomes in our diverse population of patients in our quaternary medical system which includes a largely inner city, lower income, multi-ethnic population with a high proportion of Hispanic and black patients.

Current local protocol calls for risk stratification of patients based on a modified version of the HEART Score in conjunction with serial 4th generation troponin measurements, at a 3 hour interval. Patients who have scores ≤ 3 are discharged with close outpatient follow up.

Starting data collection while the current 4th-generation troponin assay is still being used will enable us to perform a prospective, observational study on the impact of the 5th Gen Tn assay on patient throughput in the Emergency Department (ED). In particular the investigators would want to measure impact of the new assay on the amount of time it takes to evaluate a patient in the ED, as they anticipate the 5th Gen Tn will allow more rapid decision making in the clinical environment. The primary outcomes will be the change in the time it takes to make a clinical decision regarding admission or discharge to the hospital in patients presenting with possible ACS. This time interval is often referred to as the 'doctor to disposition time' or 'provider to decision time'. The investigators will also be able to evaluate impact on other throughput related factors such as admission rates.

Enrolling patients from the ED, the investigators will perform telephone follow-up 30 and 90 days following their ED visit to ascertain clinical outcomes. They will assess for any differences in the rate of major adverse cardiac events (MACE) - defined as likely cardiac death, non-fatal myocardial infarction, malignant dysrhythmia, or emergent revascularization procedures - between patients evaluated with the 4th-generation and 5th Gen Tn can be quantified, both in the discharged and admitted groups. This study will be uniquely qualified to evaluate these outcomes in a Hispanic cohort, which has been relatively underrepresented in the literature to date.

In addition, studying the new assay in a real world clinical practice will allow investigators to better understand how to interpret rapid changes in troponin values that remain below the 99th percentile normal range (14 ng/L in females, 22 ng/L in males). Multiple studies have demonstrated the utility of measuring the change in serum troponin concentration (delta-troponin) over pre-defined time intervals for identifying patients at risk for acute myocardial infarction (AMI) and MACE. In many EDs, however, limited clinical resources makes it difficult to obtain repeat blood tests on strict time frames. In the very high volume setting of the Columbia University Irving Medical Center (CUIMC) ED, the investigators expect to be able to evaluate the utility of tracking the rate of change of the 5th Gen Tn assay over multiple time points.

Being able to quantify the impact of the new test on practice patterns and ED patient throughput is critical to understanding how to best implement 5th Gen Tn into protocols that provide safe and efficient care. This data will also be of high significance not just to our local institution but to many other acute care settings and health systems across the United States as they in turn adopt this new assay over the next several years. Finally, studying this new assay in the particular socioeconomic and racial/ethnic patient mix of our institution will help understand the best way to implement this test throughout the Western hemisphere.

ELIGIBILITY:
Inclusion Criteria:

- All patients presenting to the Adult Emergency Department (age 20 and above) for whom a troponin enzyme test is collected for the purpose of evaluating for possible acute coronary syndrome.

Exclusion Criteria:

* Not fluent in English or Spanish
* Inability to participate in follow-up (incarceration, lack of telephone access, cognitive impairment, etc.)
* Patients in or immediately post cardiac arrest
* Prior heart transplant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to a single high volume, urban, tertiary care Emergency Department that sees greater than 94,000 patient visits a year in a predominantly Hispanic population.
Sampling Method: Probability Sample
Enrollment: 1949 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
ED Provider to Decision Time (ED PTDT) | Duration of index Emergency Department Visit
  Time in minutes from initial provider contact in the Emergency Department to disposition (admission versus discharge) decision.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 30 Days and 60 Days after initial Emergency Department Visit
  Incidence of likely cardiac death, myocardial infarction, malignant dysrhythmia, or emergent revascularization procedures after discharge from the ED.

CONTACTS AND LOCATIONS:
Overall Officials: Edward H. Suh, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No